CLINICAL TRIAL: NCT03188965
Title: An Open-label, First-in-human, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Maximum Tolerated Dose and / or Recommended Phase II Dose of the ATR Inhibitor BAY1895344 in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: First-in-human Study of ATR Inhibitor BAY1895344 in Patients With Advanced Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18594; 2016-004484-39 (EudraCT Number)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor; Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
Keywords: First in human; Solid tumors; Lymphomas; Dose escalation; Dose expansion
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma | interventions — BAY 1895344

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: single-agent dose-escalation (Experimental): Patients with histologically confirmed solid tumors or non-Hodgkin's lymphoma (NHL) receive BAY1895344 in a 21-day cycle.
  Interventions: Drug: Elimusertib (BAY1895344)
- Part A.1: Single-agent dose escalation with alternative dosing schedule (Experimental): Patients with histologically confirmed solid tumors or NHL known to be positive for ATM loss and/or ATM deleterious mutations receive BAY1895344 in a 28-day cycle.
  Interventions: Drug: Elimusertib (BAY1895344)
- J-arm of Part A: dose escalation cohort in Japanese patients (Experimental): Japanese patients with histologically confirmed solid tumors receive BAY1895344 at two dose levels: MTD-1 and MTD.
  Interventions: Drug: Elimusertib (BAY1895344)
- Part B: single-agent expansion (Experimental): Patients with a) DDR deficiency biomarker-positive advanced solid tumors: castration-resistant prostate cancer (CRPC), HER2-negative breast cancer (BC), colorectal cancer (CRC), and gynecological tumors; OR b) histologically confirmed advanced cancer and loss of ATM regardless of the cancer type receive BAY1895344 at MTD determined at the end of dose escalation.
  Interventions: Drug: Elimusertib (BAY1895344)
- Part B.1: single-agent expansion with alternative dosing schedule (Experimental): Patients with histologically confirmed relapsed or refractory MCL receive BAY1895344 at a dose determined after evaluation of multiple BAY1895344 doses in Part A.1
  Interventions: Drug: Elimusertib (BAY1895344)

INTERVENTIONS:
Drug: Elimusertib (BAY1895344) — Solution or tablet, oral, to be administered until evidence of tumor progression, unacceptable toxicity, consent withdrawal, or withdrawal from the study at the discretion of the investigator.

SUMMARY:
The ATR (ataxia-telangiectasia and Rad3 related protein) inhibitor BAY1895344 is developed for the treatment of patients with advanced solid tumors and lymphomas. The purpose of the proposed trial is to evaluate the safety and tolerability of BAY1895344, and to identify the maximum tolerated dose of BAY1895344 that could be safely given to cancer patients. Further, the response of the cancer to the treatment will be determined.

ELIGIBILITY:
Inclusion Criteria:

Part A - single-agent dose-escalation:

- Patients with histologically confirmed solid tumors or NHL. Patients with tumors known to be positive for deoxyribonucleic acid damage repair (DDR) defects (such as ataxia-telangiectasia mutated [ATM] deleterious mutation or low ATM expression) can be included.

J-arm of Part A - single-agent dose-escalation in Japanese:

- Japanese patients with histologically confirmed solid tumors. Patients with tumors known to be positive for DDR defects (such as ATM deleterious mutation or low ATM expression) can be included.

Part A.1 - single-agent dose-escalation with alternative dosing schedule:

- Patients with histologically confirmed solid tumors or NHL known to be positive for ATM loss and/or ATM deleterious mutations will be included. The biomarker status of patients in Part A.1 will be evaluated before general screening and only patients with the presence of the putative biomarkers of DDR deficiency will be recruited into general screening.

Part B - single-agent expansion:

* Patients with DDR deficiency biomarker-positive advanced solid tumors of the following histologies: i) CRPC; ii) HER2-negative BC that is hormone-receptor positive (estrogen-receptor positive, progesterone-receptor positive, or both) or TNBC; iii) CRC, and iv) gynecological tumors (ovarian, primary peritoneal, and fallopian tube cancers, endometrial cancer, or cervical cancer).
* Patients with histologically confirmed advanced solid cancer, regardless of the cancer type, or NHL and loss of ATM protein by IHC.
* The biomarker status of patients in Part B will be evaluated before general screening and only patients with the presence of the putative biomarkers of DDR deficiency will be recruited into general screening.

Part A.1 And Part B:

- Patients must be able to provide either samples of archival tumor tissue not older than 6 months or a fresh tumor biopsy during general screening.

Part B.1 - single-agent expansion with alternative dosing schedule:

- Patients with histologically confirmed R/R MCL. These patients do not undergo biomarker testing to determine eligibility. The provision of baseline tumor tissue (archival or fresh) is strongly encouraged. If archival tissue ≤ 6 months old is unavailable, a fresh baseline biopsy may be obtained if safe and feasible.

The following inclusion criteria apply to ALL (dose-escalation and expansion) patients:

* Patients with tumors resistant or refractory to standard treatment and in which, in the opinion of the investigator, experimental treatment with BAY1895344 may be of benefit. Furthermore, no standard therapy would confer clinical benefit to the patient. Patients in the MCL cohort of Part B.1 are to be relapsed or refractory to standard treatments.
* Patients must have measurable disease (as per Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1] or the Lugano classification as applicable, with the exception of prostate cancer patients who must have measurable or evaluable disease per the recommendations of the Prostate Cancer Clinical Trial Working Group 3 [PCWG3]).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. For MCL patients: ECOG of 0 to 2.
* Patients must have adequate bone marrow function as assessed by the following laboratory tests to be conducted within 7 (+2) days before the first dose of study drug. Note that the below values are to be independent of red blood cell transfusions or granulocytes colony-stimulating factor (G-CSF) (i.e., no red blood cell or platelets transfusion within 28 days prior to the screening complete blood count [CBC] result, or administration of G-CSF is to occur within 14 days prior to the CBC result). Requirements for MCL patients are indicated below.

  * a. Hemoglobin ≥ 9 g/dL. Patients with chronic erythropoietin treatment consistent with institutional guidelines can be included. For MCL patients: ≥ 8 g/dL; red blood cell transfusions during the screening period are allowed, and patients with chronic erythropoietin treatment consistent with institutional guidelines can be included
  * b. Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L (≥ 1500/mm^3). For MCL patients: ANC ≥ 1.0 X 10^9/L. Patients with ANC ≤ 1.0 X 10^9/L due to marrow infiltration may receive G-CSF during screening to bring pretreatment ANC levels to ≥ 1.0 X 10^9/L
  * c. Platelet count ≥ 100 X 10^9/L (≥100,000/mm^3). For MCL patients: ≥ 75 X 10^9/L

Exclusion Criteria:

* Known hypersensitivity to the study drugs or excipients of the preparations or any agent given in association with this study
* History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class >II, unstable angina (angina symptoms at rest), new-onset angina (within the past 6 months before study entry), myocardial infarction within the past 6 months before study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers, calcium channel blockers, and digoxin are permitted)
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C
* Known human immunodeficiency virus (HIV)-infected persons are not eligible if any of the following criteria apply：

  * CD4+ T-cell count less than 350 cells/μL
  * History of AIDS-defining opportunistic infection within the past 12 months
  * On established antiretroviral therapy (ART) for less than 4 weeks or presenting with a viral load of more than 400 copies/mL prior to enrollment
  * On ART or prophylactic antimicrobials that are expected to cause significant drug-drug interactions or overlapping toxicities with study intervention
* Patients who have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment. Patients with chronic HBV or HCV infection are eligible at the investigator's discretion provided that the disease is stable and sufficiently controlled under treatment.
* Infections of Common Terminology Criteria for Adverse Events Version (CTCAE) Grade 2 not responding to therapy or active clinically serious infections of CTCAE Grade > 2
* Metastatic solid brain, spinal, or meningeal tumors or central nervous system (CNS) lymphoma manifestations (including meningeosis lymphomatosa and parenchymal lymphoma lesions) unless the patient is > 3 months from definitive therapy, has a stable imaging study within 4 weeks prior to the first dose of study drug and is clinically stable with respect to the tumor at the time of study entry. Patients with asymptomatic brain metastases must not be on steroid therapy. Patients with neurological symptoms should undergo a CT / MRI scan of the brain or spinal column to exclude new or progressive brain, meningeal, or spinal metastases or CNS lymphoma manifestations.
* History of organ allograft transplantation. For MCL patients: Those who received an allogeneic stem cell transplant may participate provided that engraftment has occurred, there is no evidence of GVHD, and the patient is not taking immune suppressants. MCL patients who received an autologous stem cell transplant may participate once they have recovered from the procedure.
* Treatment with anticancer chemotherapy or immunotherapy during the study or within 3 weeks before the first dose of study drug. For small-molecule drugs, a period of at least 3 half-lives before the first dose of study drug is acceptable. Mitomycin C or nitrosoureas should not be given within 6 weeks before the first dose of study drug.
* Treatment with systemic steroids (methylprednisolone dose ≥10 mg/day or equivalent dose). For MCL patients: Treatment with systemic corticosteroids > 20 mg/day prednisone equivalent (unless patient has been taking a stable dose for >3 weeks and has shown tumor progression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) and / or recommended Phase II dose (RP2D) of BAY1895344 | Up to 6 months, minimum: 1 cycle (= 21days)
  MTD and/or R2PD will be determined in Cycle 1 of Part A, Part A.1 and J-arm of Part A.
  The MTD is defined as the maximum dose at which the incidence of dose-limiting toxicities (DLTs) during Cycle 1 is below 30%, or the maximum dose tested, whichever is achieved first during dose-escalation.
Incidence of DLTs during Cycle 1 in dose-escalation cohorts during Part A of the study | During Cycle 1, 1 cycle=21 days
Incidence of DLTs during Cycle 1 in dose-escalation cohorts during Part A.1 of the study | During Cycle 1, 1 cycle=28 days
Incidence of DLTs during Cycle 1 in dose-escalation cohorts during J-arm of the study | During Cycle 1, 1 cycle=21 days
The incidence of serious and nonserious treatment-emergent adverse events (TEAEs) | After first administration of study drug up to 30 days after the last dose of study drug
Area under the plasma concentration of BAY1895344 vs. time curve from zero to 12 hours after single-dose (AUC[0-12]) and multiple-dose administrations (AUC[0-12]md) in Cycle 1 | Pre-dose and up to 12 hours post-dose at Day 1 of Cycle 1 and Day 10 (Part A and J-arm) or Day 17 (Part A.1) of Cycle 1
  AUC(0-12) and AUC(0-12)md will be evaluated in Part A, A.1 and J-arm of Part A.
Maximum observed drug concentration in plasma of BAY1895344 after single-dose (Cmax) and multiple-dose administrations (Cmax,md) in Cycle 1 | Pre-dose and up to 12 hours post-dose at Day 1 of Cycle 1 and Day 10 (Part A and J-arm) or Day 17 (Part A.1) of Cycle 1
  Cmax and Cmax,md will be evaluated in Part A, A.1 and J-arm of Part A.

SECONDARY OUTCOMES:
Incidence of solid tumor responses (except CRPC) consistent with the RECIST 1.1 criteria | Through study completion, an average of 4 months
  Responses include: CR (complete response), PR (partial response), SD (stable disease), PD (progressive disease). CRPC: castration resistant prostate cancer; RECIST: Response Evaluation Criteria in Solid Tumors
Incidence of lymphoma responses consistent with the Lugano Classification | Through study completion, an average of 4 months
  Responses include: CR (complete response), PR (partial response), SD (stable disease), PD (progressive disease).
Incidence of CRPC tumor responses consistent with the recommendations of the PCWG3 | Through study completion, an average of 4 months
  Responses include: CR (complete response), PR (partial response), SD (stable disease), PD (progressive disease).
  PCWG3: Prostate Cancer Working Group 3

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- United States (14):
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - US Oncology / Eugene, Eugene, Oregon
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology- San Antonio Northeast, San Antonio, Texas
  - University of Utah - Oncology, Salt Lake City, Utah
  - Fairfax-Northern Virginia Hematology/Oncology, PC, Fairfax, Virginia
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - OHRI - The Ottawa Hospital, Ottawa, Ontario
  - Integrated Cancer Center of the CHU de Québec, Québec
- Beijing Cancer Hospital, Beijing, China
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Center Singapore, Singapore
- Switzerland (3):
  - Hôpital Cantonal Universitaire de Genève, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Oncology Institute of Southern Switzerland, Bellinzona
- United Kingdom (3):
  - Velindre Hospital, Cardiff, South Glamorgan
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Lucking U, Wortmann L, Wengner AM, Lefranc J, Lienau P, Briem H, Siemeister G, Bomer U, Denner K, Schafer M, Koppitz M, Eis K, Bartels F, Bader B, Bone W, Moosmayer D, Holton SJ, Eberspacher U, Grudzinska-Goebel J, Schatz C, Deeg G, Mumberg D, von Nussbaum F. Damage Incorporated: Discovery of the Potent, Highly Selective, Orally Available ATR Inhibitor BAY 1895344 with Favorable Pharmacokinetic Properties and Promising Efficacy in Monotherapy and in Combination Treatments in Preclinical Tumor Models. J Med Chem. 2020 Jul 9;63(13):7293-7325. doi: 10.1021/acs.jmedchem.0c00369. Epub 2020 Jun 28. PMID 32502336